CLINICAL TRIAL: NCT04423731
Title: Neoadjuvant Chemotherapy in Borderline Resectable and Locally Advanced Pancreatic Cancer - a Norwegian Population Based Observational Study (NORPACT-2)
Brief Title: Neoadjuvant Chemotherapy in Borderline Resectable and Locally Advanced Pancreatic Cancer (NORPACT-2)
Status: Active, not recruiting | Type: Observational
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Knut Jørgen Labori, Consultant surgeon MD, PhD, Oslo University Hospital
Other Study IDs: 2017/1382/REK nord
Record Dates: First submitted 2020-06-04; First posted 2020-06-09 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Locally Advanced Pancreatic Adenocarcinoma; Chemotherapy Effect; Borderline Resectable Pancreatic Adenocarcinoma; Pancreatectomy
MeSH Terms: interventions — folfirinox; Gemcitabine; Fluorouracil; Leucovorin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Folfirinox — Neoadjuvant chemotherapy is given according to different regimens, preferably FOLFIRINOX according to the recommendations in the national Norwegian guidelines. The choice of chemotherapy regimen is decided by the treating oncologist.
  Other Names: Gemcitabine/nab-paclitaxel; Gemcitabine; 5-FU (fluorouracil) and leucovorin; FLOX

SUMMARY:
This is a Norwegian prospective observational study that evaluates the resectability rate in patients with borderline resectable and locally advanced pancreatic cancer who received neoadjuvant chemotherapy in a population based cohort. Eligible patients are treated with neoadjuvant chemotherapy possibly followed by surgical exploration and resection. All Norwegian centres performing pancreatic surgery have agreed to collaborate in this trial. The assignment of the medical intervention is not at the discretion of the investigator, but follow the national Norwegian guidelines regarding diagnostic work up, oncological and surgical treatment and follow up.

ELIGIBILITY:
Inclusion Criteria:

* borderline resectable or locally advanced adenocarcinoma of the pancreas (NCCN, version 2, 2015)
* Nx, M0 (UICC 8 th version, 2016)
* cytological or histological confirmation of adenocarcinoma
* age > 18 year and considered fit for major surgery
* written informed consent
* considered able to receive the study-specific chemotherapy

Exclusion Criteria:

* co-morbidity precluding pancreatectomy
* chronic neuropathy ≥ grade 2
* WHO performance score > 2
* granulocyte count < 1500 per cubic millimetre
* platelet count < 100 000 per cubic millimetre
* serum creatinine > 1.5 UNL (upper limit normal range)
* albumin < 2,5 g/dl
* female patients in child-bearing age not using adequate contraception, pregnant or lactating women
* mental or physical disorders that could interfere with treatment of with the provision of informed consent
* any reason why, in the opinion of the investigator, the patient should not participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Population based cohort from a universal health care system
Sampling Method: Non-Probability Sample
Enrollment: 251 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of resectability in both groups (borderline and locally advanced pancreatic cancer) | 5 years
  Patients who undergo surgical resection will be documented

SECONDARY OUTCOMES:
Overall survival from time of inclusion (intention to treat) | Overall survival rate at 5 years using Kaplan-Meier survival analysis
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 1 year after inclusion
Overall survival following resection | Overall survival rate at 5 years using Kaplan-Meier survival analysis
Overall survival after 1, 2, 3 and 5 years | 1, 2, 3 and 5 years after inclusion
1-year progression-free survival rate | 1-year after surgical resection
Disease-free survival | Disease-free survival at 5 years using Kaplan-Meier survival analysis
Radiological response | 2-6 months after initiation of chemotherapy
Histopathological response | 14-30 days post surgery
R0 resection rate | 14-30 days post surgery
Complication rates after surgery classification systems) | 30 and 90 days post surgery
  Dindo-Clavien and ISPGS
Completion rates of all parts of multimodal treatment | Up to 1 year after inclusion
QoL (EORTC QLQ-30) | 5 years
Performance status - Eastern Cooperative Oncology Group (ECOG) | 5 years
  0 - Asymptomatic (Fully active, able to carry on all predisease activities without restriction)
  1. - Symptomatic but completely ambulatory (Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature. For example, light housework, office work)
  2. - Symptomatic, <50% in bed during the day (Ambulatory and capable of all self care but unable to carry out any work activities. Up and about more than 50% of waking hours)
  3. - Symptomatic, >50% in bed, but not bedbound (Capable of only limited self-care, confined to bed or chair 50% or more of waking hours)
  4. - Bedbound (Completely disabled. Cannot carry on any self-care. Totally confined to bed or chair)

CONTACTS AND LOCATIONS:
Overall Officials: Knut J. Labori, MD, PhD, Principal Investigator — Oslo University Hospital, Oslo, Norway
Locations (1):
- Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Farnes I, Lund-Iversen M, Aabakken L, Verbeke C, Labori KJ. Molecular testing for personalized therapy is underutilized in patients with borderline resectable and locally advanced pancreatic cancer - real world data from the NORPACT-2 study. Scand J Gastroenterol. 2024 Sep;59(9):1093-1096. doi: 10.1080/00365521.2024.2373115. Epub 2024 Jul 3. PMID 38957079
- [Background] Farnes I, Paulsen V, Verbeke CS, Tonnesen CJ, Aabakken L, Labori KJ. Performance and safety of diagnostic EUS FNA/FNB and therapeutic ERCP in patients with borderline resectable and locally advanced pancreatic cancer - results from a population-based, prospective cohort study. Scand J Gastroenterol. 2024 Apr;59(4):496-502. doi: 10.1080/00365521.2023.2290456. Epub 2023 Dec 21. PMID 38126766
- [Background] Farnes I, Kleive D, Verbeke CS, Aabakken L, Issa-Epe A, Smastuen MC, Fosby BV, Dueland S, Line PD, Labori KJ. Resection rates and intention-to-treat outcomes in borderline and locally advanced pancreatic cancer: real-world data from a population-based, prospective cohort study (NORPACT-2). BJS Open. 2023 Nov 1;7(6):zrad137. doi: 10.1093/bjsopen/zrad137. PMID 38155512